CLINICAL TRIAL: NCT01881243
Title: Reoxygenation After Cardiac Arrest (REOX Study)
Acronym: REOX
Status: Completed | Type: Observational
Sponsor: The Cooper Health System (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: REOX; R01HL112815 (NIH)
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Cardiac Arrest
Keywords: Cardiac Arrest, Hyperoxia, Ischemia-reperfusion Injury, Reactive Oxygen Species, Oxidative Stress, Neuropsychological Tests
MeSH Terms: conditions — Heart Arrest; Hyperoxia; Reperfusion Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This research will measure biomarkers of oxidative stress (isoprostanes and isofurans) on plasma samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult patients resuscitated from cardiac arrest

SUMMARY:
The broad objective of this study is to test the association between hyperoxia exposure after resuscitation from cardiac arrest and outcome. Our overarching hypothesis is that hyperoxia after ROSC is associated with increased oxidative stress and worsened neurological and cognitive outcomes.

DETAILED DESCRIPTION:
Specific Aim 1: Test if the degree and duration of hyperoxia following ROSC from cardiac arrest is associated with the degree of in vivo oxidative stress during the post-resuscitation phase of therapy.

Approach: We will conduct a multicenter prospective observational study of adult patients resuscitated from cardiac arrest. We will record data pertaining to oxygenation parameters and other factors and measure biomarkers of oxidative stress (isoprostanes and isofurans) in the plasma at 0 and 6 hours after ROSC using gas chromatography negative ion chemical ionization mass spectrometry. We will determine the exposure to post-ROSC hyperoxia by calculating the time-weighted average PaO2 and SaO2 for the post-resuscitation phase of therapy, and will test the association with plasma isoprostane and isofuran levels.

Specific Aim 2: Test if the degree and duration of hyperoxia following ROSC from cardiac arrest is associated with the degree of neurological disability at hospital discharge.

Approach: In the study described above, we will determine the Modified Rankin Scale at hospital discharge. We will perform multivariable analyses adjusted for numerous covariates known to be associated with outcome in post-cardiac arrest patients to determine if post-ROSC hyperoxia exposure is independently associated with neurological disability.

Specific Aim 3: Test if the degree and duration of hyperoxia following ROSC from cardiac arrest is associated with neuropsychological outcomes among survivors at 180 days.

Approach: In the study described above, we will assess neuropsychological outcome among survivors at 180 days. Neuropsychological testing will use validated instruments across five cognitive domains (attention, Wechsler Adult Intelligence Scale-IV-digit span; (2) reasoning, Wechsler Adult Intelligence Scale-IV-similarities; (3) immediate and delayed memory, Wechsler Memory Scale-III-logical memory I and II; (4) verbal fluency, Controlled Oral Word Association Test; and (5) executive functioning, Hayling Sentence Completion Test). We will perform multivariable analyses to determine if post-ROSC hyperoxia exposure is independently associated with neuropsychological deficits.

ELIGIBILITY:
Inclusion Criteria:

* Age >17 years
* Cardiac arrest
* Return of spontaneous circulation
* Not following commands immediately after ROSC
* Endotracheal intubation
* Clinician intent to treat with therapeutic hypothermia (or absence of clinician intent to withhold therapeutic hypothermia)

Exclusion Criteria:

* Presumed etiology of arrest is trauma
* Presumed etiology of arrest is hemorrhage
* Presumed etiology of arrest is sepsis
* Permanent resident of nursing home or other long-term care facility
* Any other condition, that in the opinion of the investigator, would preclude the subject from being a suitable candidate, e.g. end stage chronic illness with no reasonable expectation of survival to hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients resuscitated from cardiac arrest
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2013-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Plasma isoprostanes/isofurans (mechanistic outcome) | 0 and 6 hours post-ROSC

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) (primary neurological outcome) | hospital discharge

OTHER OUTCOMES:
Cognitive testing (primary neuropsychological outcome) | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Trzeciak, MD, MPH, Study Director — The Cooper Health System
Locations (5):
- United States (5):
  - Indiana University/ Methodist Hospital, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cooper University Hospital, Camden, New Jersey
  - Hospital of the University of Pennsylvania and Penn Presbyterian Medical Center, Philadelphia, Pennsylvania